CLINICAL TRIAL: NCT07269314
Title: Introduzione Della Polymerase Chain Reaction (PCR) in Microbiologia e Parassitologia
Brief Title: Introduction of Polymerase Chain Reaction (PCR) in Microbiology and Parasitology
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefania Paolucci, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: P_41
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Malaria, Pneumocystis, Leishmania
MeSH Terms: conditions — Malaria; Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal is to develop molecular systems to support or replace in microscopic characterization and in vitro tests with molecular biology systems capable of improving performance in parasitology tests. In particular, we will analyze the main pathogens: several Leishmania species (Old and New World Leishmania species), the five Plasmodium species of human interest (falciparum, oval, vivax, malariae and knowlesi) and Pneumocistys jiroveci, using molecular methods based on the speed, specificity and sensitivity necessary for their diagnosis. Furthermore, we want to provide specific elements for the typing of the species. Our aim is to improve diagnostic and specie classification methods by using PCR in microbiology and parasitology, to evaluate its impact on diagnosis. We would evaluate the impact of this method in terms of timing, sensitivity and specificity of diagnosis. We would also explore future possibilities on quantification techniques, in order to support the clinician to evaluate the efficacy of therapy during the follow-up.

Furthermore, we would evaluate these methods in terms of cost effectiveness towards classical direct methods, which are now operator-dependent.

DETAILED DESCRIPTION:
Our project is an observational retrospective and prospective cross-sectional diagnostic pilot study, about the comparison between standard routine laboratory tests and new molecular biology assays. In particular, we would detect principal pathogen Leishmania species (Old and New World Leishmania species), the five species of Plasmodium of human interest (falciparum, oval, vivax, malaria and knowlesi) and Pneumocistys jiroveci,

1. Positive samples for Leishmania amastygotes in peripheral blood and/or bone marrow aspirate/biopsy and/or from cutaneous scraping/biopsy previously tested according to routine diagnostic assays will be tested with a specific qualitative PCR analysis by using commercial diagnosis kit. In addition, we would perform a system of DNA quantification using PCR cycle threshold of the single sample and a virtual scale able to convert the results in the DNA load (Piralla A et al, J clin virol 2013). Then we would perform a specific DNA sequencing of p70 gene to determine specie and the strain.
2. Plasmodium species blood positive samples tested for and analyzed by direct microscopy and immunocromatographic assay, will be tested with multiplex PCR commercial diagnostic kit or with a described method (A.Berg et al, Infection 2020) able to determine single or mixed infection and to quantify the parasitemia respectively. In detail, the blood samples will be analyzed with qualitative and quantitative PCR analysis for Plasmodium spp and Plasmodium Falciparum, respectively. The concentration of P. falciparum DNA in blood samples will be measured by quantitative real-time PCR (qPCR) as described elsewhere (Imwong M, J.clin.microb 2014). In Plasmodium falciparum positive samples, the amount of DNA copies obtained from each sample will be compared with the level of parasitemia obtained from direct microscopy analysis. In this way we would like to determine a range of DNA copy values comparable to the different degrees of classification that are currently obtained with percentages of red blood cells positive for the infection (<5% vs >5%). In this way, it could be possible to assess a level of parasitemia with quantitative PCR techniques.
3. Finally, detection of Pneumocistis jirovecii in positive BAL or bronchoaspirate (BAS) samples obtained by direct microscopy will be reanalyzed by using PCR commercial diagnostic kit. As previously mentioned, the CT value will be converted in DNA load in comparison with direct microscopy data.

ELIGIBILITY:
Inclusion Criteria:

Approximately 200-300 samples retrospectively submitted to the laboratory for the study in question, for the detection of P. jirovecii, Plasmodium Malaria and Leishmania tested with the classical method.

Exclusion Criteria:

Samples that are unsuitable due to storage errors and/or insufficient volume will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Positive samples for Leishmania amastygotes in peripheral blood and/or bone marrow aspirate/biopsy and/or from cutaneous scraping/biopsy previously tested according to routine diagnostic assays 2-Plasmodium species blood positive samples tested for and analyzed by direct microscopy and immunocromatographic assay, 3-Pneumocistis jirovecii in positive BAL or bronchoaspirate (BAS) samples obtained by direct microscopy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pneumocystis PCR test | From January 2024 to september 2025
  Primary endpoint will be the estimation of sensitivity of PCR tests in identifying the presence of main pathogens: Leishmania species, Plasmodium species and Pneumocistys jiroveci.

SECONDARY OUTCOMES:
Malaria PCR test | From genuary 2025 to september 2026
  Secondary endpoint will be the comparison of the concentration of P. falciparum DNA in blood samples (measured by qPCR) according to parasitemia (>5% vs <5%).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No